CLINICAL TRIAL: NCT07020104
Title: The Role of Skin Sodium Accumulation in Chronic Kidney Disease
Acronym: SKIN-CKD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Dutch Kidney Foundation (Other)
Responsible Party: Principal Investigator, Rik Olde Engberink, Internist-nephrologist, clinical pharmacologist, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NL82810.018.22
Record Dates: First submitted 2025-04-15; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Diseases
Keywords: Skin sodium; Sodium MRI; CKD; Prognosis; Cardiovascular event; Renal event; Quality of life; Tissue sodium
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Hydrochlorothiazide; Spironolactone; lercanidipine

STUDY DESIGN:
Intervention Model Description: The association between tissue sodium accumulation and cardiovascular parameters, body composition, skin hydration and transepidermal water loss, renal and cardiovascular outcome will be studied in 60 CKD patients (A).
  14 of the 60 CKD patients will be randomized to a 2-week low sodium diet and a 2-week high sodium diet in an open-label cross-over manner (B).
  12 CKD patients will receive 3 antihypertensive agents (spironolactone, lercanidipine and hydrochlorothiazide) in random order for 6 weeks (C).
  12 of the 60 CKD subjects will be randomized to a 4 week increased water intake and 4 week habitual water intake (D).
  All the intervention mentioned above are separated by a washout period of at least 2 weeks between interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sodium excretion intervention (C) (Experimental): In this intervention group, the patients will receive three antihypertensive drugs in a randomized order. Thus the following orders are possible:
  1. Lercanidipine - Spironolactone - Hydrochlorothiazide
  2. Lercanidipine - Hydrochlorothiazide - Spironolactone
  3. Hydrochlorothiazide - Lercanidipine - Spironolactone
  4. Hydrochlorothiazide - Spironolactone - Lercanidipine
  5. Spironolactone - Lercanidipine - Hydrochlorothiazide
  6. Spironolactone - Hydrochlorothiazide- Lercanidipine
  Interventions: Drug: Hydrochlorothiazide; Drug: Spironolactone; Drug: Lercanidipine
- Sodium intake intervention (B) (Experimental): In this intervention group, the patients will receive two sodium diets in a randomized order. The following orders are possible:
  1. High sodium intake- Low sodium intake
  2. Low sodium intake- High sodium intake
  Interventions: Dietary Supplement: High sodium dietary intake (>200mmol/l); Dietary Supplement: Low sodium dietary intake (<50mmol/l)
- Water intake intervention (D) (Experimental): In this intervention group, the patients will be prescribed two water interventions in a randomized order. The following orders are possible: 1. High water intake- Habitual water intake 2. Habitual water intake- High water intake
  Interventions: Dietary Supplement: High water intake; Dietary Supplement: Habitual water intake

INTERVENTIONS:
Drug: Hydrochlorothiazide — Each patient will receive 1 tablet of hydrochlorothiazide 12.5mg once a day for the first 3 weeks of the drug cycle. If clinical and biochemical parameters allow, the dosage is doubled to 2 tablets of hydrochlorothiazide 12.5mg once daily for the following 3 weeks.
  If the laboratory results and clinical parameters do not allow dose intensification, the initial dosage will be continued during the second half of the drug cycle.
  Arms: Sodium excretion intervention (C)
Drug: Spironolactone — Each patient will receive 1 tablet of spironolacton 12.5mg once a day for the first 3 weeks of the drug cycle. If clinical and biochemical parameters allow, the dose is doubled to 2 tablets of spironolacton 12.5mg once daily for the following 3 weeks.
  If the laboratory results and clinical parameters do not allow dose intensification, the initial dosage will be continued during the second half of the drug cycle.
  Arms: Sodium excretion intervention (C)
Drug: Lercanidipine — Each patients will receive 1 tablet of lercanidipine 10mg once a day for the first 3 weeks of the drug cycle. If clinical and biochemical parameters allow, the dose is doubled to 2 tablets of lercanidipine 10mg once daily for the following 3 weeks.
  If the laboratory results and clinical parameters do not allow dose intensification, the initial dosage will be continued during the second half of the drug cycle.
  Arms: Sodium excretion intervention (C)
Dietary Supplement: High sodium dietary intake (>200mmol/l) — The patients will receive a 2-week high sodium diet. The patients will receive dietary advice to achieve this goal of >200mmol/l sodium (>12g salt) intake per day.
  Arms: Sodium intake intervention (B)
Dietary Supplement: Low sodium dietary intake (<50mmol/l) — The patients will receive a 2-week low sodium diet. The patients will receive dietary advice to achieve this goal of <50mmol/l sodium (<3g salt) intake per day.
  Arms: Sodium intake intervention (B)
Dietary Supplement: High water intake — During the increased water intake period, the patients will be instructed to drink 1 L more than their mean 24-hour urine volume at screening and baseline.
  Arms: Water intake intervention (D)
Dietary Supplement: Habitual water intake — During this part of the intervention, the patients will be instructed to maintain their habitual water intake.
  Arms: Water intake intervention (D)

SUMMARY:
This project consists of four substudies: a cohort study (A) and a sodium intake intervention (B) and a sodium excretion intervention (C) and a water intervention study (D).

The main objective of the cohort study (A) is to investigate the prognostic implications of tissue sodium accumulation in CKD patients. The primary objective of the sodium intervention studies is to study the effect of high and low sodium intake (B) and increased renal sodium excretion (C) on tissue sodium content. The main objective of the water intervention study (D) is to investigate the effect of increased and habitual water intake on tissue sodium content and transepidermal water loss.

DETAILED DESCRIPTION:
Cohort study (A):

60 CKD patients (eGFR 15 - 60 ml/min/1.73m2) are included in this cohort study. At the start of the study the association between tissue sodium content and micro-and macrovascular function will be evaluated. These patients will be followed up to investigate the association between tissue sodium content, quality of life and renal and cardiovascular events.

Sodium intake intervention (B):

A subgroup of 14 CKD patients (eGFR 15 - 60 ml/min/1.73m2) will be randomized to a 2-week low sodium diet and a 2-week high sodium diet in a cross-over study.

Sodium excretion intervention (C):

A subgroup of 12 CKD patients (eGFR 30 - 60 ml/min/1.73m2) with hypertension will be randomized to receive 6 weeks of treatment with hydrochlorothiazide, spironolactone and lercanidipine in a randomized open-label cross-over trial.

Water intake intervention (D) A subgroup of 12 CKD patients (with eGFR 15-30 ml/min/1.73m2, hypertension and fasting morning urine osmolality < 425 mOsm/kg for men and < 400 mOsm/kg for women) will be randomized to a 4-week habitual water intake and 4-week increased water intake in a cross-over study.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic kidney disease with an eGFR between 15 and 60 ml/min/1.73m2.
2. Stable diuretic and antihypertensive treatment for the previous 6 weeks.

Additional inclusion criteria for the sodium excretion intervention 1. Office systolic blood pressure (SBP) >135 mmHg

Additional inclusion criteria for the water intervention

1. Chronic kidney disease with an eGFR between 15 and 29 ml/min/1.73m2
2. Office blood pressure ≥140/90 mmHg or use of antihypertensive medication
3. Fasting morning urine osmolality <425 mOsm/kg for men and < 400 mOsm/kg for women

Exclusion Criteria:

1. Age <18 years.
2. The patient is expected to start renal replacement therapy or is planned to receive a kidney transplantation within 3 months.
3. An active diagnosis of nephrotic syndrome at inclusion.
4. (Recurrent) acute glomerulonephritis within 1 year prior to the study.
5. Salt losing nephropathy.
6. Use of oral or intravenous glucocorticoids with an equivalent of prednisolone >5mg/day.
7. Contra-indication for MRI.
8. Cardiovascular event/ surgery in the previous 3 months.
9. Pregnant women, women of child bearing age planning to conceive for the study duration, women of child bearing age without contraception.
10. Participation in other (pharmacological) intervention studies.
11. Presence of significant comorbidities with a life expectancy of less than 1 year.
12. Disorder that compromises the participants' ability to give truly informed consent for participation in this study.
13. Patients with an active infection and/or auto-immune diseases with involvement of the lower extremities.
14. Any other issues that in opinion of the investigator could be harmful to the subject or compromise interpretation of the data.

Additional exclusion criteria for the sodium intake intervention

1. Chronic use of NSAID

Additional exclusion criteria for the sodium excretion intervention

1. Serum potassium concentration >5.0 mmol/l.
2. eGFR <30 ml/min/1.73m2
3. Uncontrolled hypertension (>180/100 mmHg)
4. Severe heart failure with left ventricular ejection fraction <30%.
5. Contra-indication for investigational drugs.
6. Severe symptoms of (orthostatic) hypotension.
7. Patients with obstruction of the outflow tract of the left ventricle such as aortic valve stenosis.
8. Refractory hypokalemia, hyponatremia or hypercalcemia.
9. Severe liver insufficiency Child Pugh B/C
10. Chronic use of NSAID.

Additional exclusion criteria for the water intake intervention

1. Recent history of severe hyponatremia (outpatient plasma sodium < 130 mmol/L in the last 6 months)
2. Plasma sodium <135 mmol/L at screening
3. History of heart failure
4. Use of lithium, vasopressin analoga, vasopressin antagonists, oral or intravenous glucocorticoids, thiazide diuretics.
5. 24-hour urine volume > 2L
6. Chronic use of NSAID

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2039-12-01 (Estimated); Study Completion 2039-12-01 (Estimated)

PRIMARY OUTCOMES:
Skin sodium content at baseline (A) | 0 week
  Skin sodium content will be measured using the 7T sodium MRI
Muscle sodium content at baseline (A) | 0 week
  Muscle sodium content will be measured using the 7T sodium MRI
Change from baseline in tissue sodium content after low and high sodium diet (B) | 2 weeks
Change in tissue sodium content after treatment with hydrochloorthiazide, spironolacton and lercanidipine (C) | 6 weeks
  To study the effect of hydrochloorthiazide, spironolacton and lercanidipine on tissue sodium content, to compare the effect among the various antihypertensive agents and to assess the effect of blood pressure regulation, increased renal sodium excretion and aldosteron blockade on tissue sodium content.
Change from baseline in tissue sodium content after habitual and high water intake (D) | 4 weeks
  To evaluate the effect of high and habitual water intake on tissue sodium content.
Change from baseline in transepidermal water loss after habitual and high water intake (D) | 4 weeks
  To evaluate the effect of high and habitual water intake on transepidermal water loss.
Incidence of hyponatremia and hypervolemia (D) | 4 weeks
  Safety of high water intake in CKD patients with eGFR between 15 and 30ml/min/1.73m2

SECONDARY OUTCOMES:
Correlation between tissue sodium content and total vessel density (A) | 0 week
  Correlation between tissue sodium content measured with 7T Na-MRI and total vessel density using Sidestream Dark Field imaging.
Correlation between tissue sodium content and perfused vessel density (A) | 0 week
  Correlation between tissue sodium content measured with 7T Na-MRI and perfused vessel density using Sidestream Dark Field imaging.
Correlation between tissue sodium content and proportion of perfused vessels (A) | 0 week
  Correlation between tissue sodium content measured with 7T Na-MRI and proportion of perfused vessels using Sidestream Dark Field imaging.
Correlation between tissue sodium content and microvascular flow index (A) | 0 week
  Correlation between tissue sodium content measured with 7T Na-MRI and microvascular flow index using Sidestream Dark Field imaging.
Correlation between tissue sodium content and microvascular health score (A) | 0 week
  Correlation between tissue sodium content measured with 7T Na-MRI and microvascular health score using Sidestream Dark Field imaging.
Correlation between tissue sodium content and total pheripheral resistance (A) | 0 week
  Total pheripheral resistance will be measured using the Nexfin device and tissue sodium content will be measured using the 7T Na-MRI
Correlation between tissue sodium content and cardiac output (A) | 0 week
  Cardiac output will be measured using the Nexfin device and tissue sodium content will be measured using the 7T Na MRI
Correlation between tissue sodium content and transepidermal water loss (A) | 0 week
  Transepidermal water loss will be measured with the Tewameter® TM Hex probe and tissue sodium content will be measured using the 7T Na MRI
Correlation between tissue sodium content and office systolic and diastolic blood pressure (A) | 0 week
  Tissue sodium content will be measured using the 7T sodium MRI
Correlation between tissue sodium content and 24-hour systolic and diastolic blood pressure (A) | 0 week
  Tissue sodium content will be measured using the 7T Na MRI
Correlation between tissue sodium content and nightime blood pressure dipping pattern (A) | 0 week
  The nighttime blood pressure dipping pattern will be measured with a 24-hour blood pressure measurements. Patients will be classified as a 'dippers' when the nighttime systolic blood pressure and/or diastolic blood pressure falls >10% and <20% compared to daytime readings. Exteme dippers are described as those with blood pressure fall of at least 20%. Patients with blood pressure fall between 0 and 10% are classified as non-dippers.
Correlation between tissue sodium content and total body water (A) | 0 week
  Total body water (liter) will be measured using the bioelectrical impendance analysis and tissue sodium content will be measured using the 7T Na MRI
Correlation between tissue sodium content and quality of life (A) | At baseline and yearly during follow-up
  Quality of life(QoL) will be measured with the Kidney Disease Quality of Life questionnaire at baseline and yearly during follow-up and tissue sodium comntent will be measured using the 7T Na MRI at baseline
The correlation between tissue sodium content and traditional cardiovascular risk factors (A) | 15 years
  In the cohort study, the correlation between tissue sodium content measured with 7T Na MRI and the known traditional cardiovascular risk factors will be studied.
Change from baseline in plasma co-peptine concentrations (D) | 4 weeks
  For waterintake intervention study
Change from baseline in seated systolic and diastolic office blood pressure (B/C/D) | 2 weeks
  Seated office systolic and diastolic blood pressure after interventions compared to baseline
Change from baseline in 24-hour systolic and diastolic blood pressure (B/C/D) | 2 weeks
  24-hour systolic and diastolic blood pressure after interventions compared to baseline
Change from baseline in percentage of patients with a night-time blood pressure dipping pattern (B/C/D) | 2 weeks
  Nighttime blood pressure dipping status will be measured with a 24-hour blood pressure measurements. Patients will be classified as a 'dippers' when the nighttime systolic blood pressure and/or diastolic blood pressure falls >10% and <20% compared to daytime readings. Exteme dippers are described as those with blood pressure fall of at least 20%. Patients with blood pressure fall between 0 and 10% are classified as non-dippers.
Change from baseline in transepidermal water loss (B/C/D) | 2 weeks
  Transepidermal water loss will be measured with the Tewameter® TM Hex probe
Change from baseline in total body water (B/C/D) | 2 weeks
  Total body water will be measured using the bioelectrical impendance analysis
Change from baseline in total vessel density (B/C/D) | 2 weeks
  The total vessel density will be measured using Sidestream Dark Field imaging.
Change from baseline in perfused vessel density (B/C/D) | 2 weeks
  The perfused vessel density will be measured using Sidestream Dark Field imaging.
Change from baseline in proportion of perfused vessel (B/C/D) | 2 weeks
  The proportion of perfused vessels will be measured using Sidestream Dark Field imaging.
Change from baseline in microvascular flow index (B/C/D) | 2 weeks
  The microvascular flow index will be measured using Sidestream Dark Field imaging.
Change from baseline in microvascular health score (B/C/D) | 2 weeks
  The microvascular health score will be measured using Sidestream Dark Field imaging.
Change from baseline in total peripheral resistance (B/C/D) | 2 weeks
  The total pheripheral resistance will be measured using the Nexfin device
Change from baseline in cardiac output (B/C/D) | 2 weeks
  The cardiac output will be measured using the Nexfin device

OTHER OUTCOMES:
Skin water content at baseline (A) | 0
  Skin water content will be measured using the 7T H-MRI
Muscle water content at baseline (A) | 0 week
  Muscle water content will be measured using the 7T H-MRI
Change from baseline in skin water content (B/C/D) | 2 weeks
  Change in skin water content after sodium excretion, sodium intake and water intake intervention
Change from baseline in muscle water content (B/C/D) | 2 weeks
  Change in muscle water content after sodium excretion, sodium intake and water intake intervention
Association between tissue sodium content and skin hydration (A) | 0 week
  The skin hydration will be measured using the Corneometer® CM 825 probe
Change from baseline in skin hydration (B/C/D) | 2 weeks
  The skin hydration will be measured using the Corneometer® CM 825 probe

CONTACTS AND LOCATIONS:
Overall Officials: Rik Olde Engberink, MD, PhD, Principal Investigator — Amsterdam UMC, location AMC
Locations (1):
- Amsterdam UMC, Amsterdam-Zuidoost, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researcher